CLINICAL TRIAL: NCT02439489
Title: Phase Ib Study of the Combination of BKM120 and Cisplatin or Carboplatin in Patients With Advanced Solid Tumors
Brief Title: Study of the Combination of BKM120 and Cisplatin or Carboplatin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-11-F01b
Record Dates: First submitted 2015-04-21; First posted 2015-05-08 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BKM120-CIS (Experimental): BKM120 (60, 80 100 mg po continuously) and Cisplatin (iv 75 mg/m2)
  Interventions: Drug: BKM120-CIS
- BKM120-CARBO (Experimental): BKM120 and (60, 80 100 mg po continuously) and Carboplatin (iv AUC 5)
  Interventions: Drug: BKM120-CARBO

INTERVENTIONS:
Drug: BKM120-CIS — BKM120 will be delivered orally once daily on continuous at the dose of 60 mg (dose level 1), 80 mg (dose level 2) and 100 (dose level 3). Cisplatin will be delivered intravenously at the dose of 75 mg/m2 on day 1 every 3 weeks at each dose level of BKM120.
  In the absence of BKM120 DLT, each level will be administered to 3 patients A minimum of 2 cycles per each dose level will be administered in the absence of disease progression or toxicity
  Other Names: Buparlisib (BKM120); CISPLATINO TEVA
  Arms: BKM120-CIS
Drug: BKM120-CARBO — BKM120 will be delivered orally once daily on continuous at the dose of 60 mg (dose level 1), 80 mg (dose level 2) and 100 (dose level 3). Carboplatin will be delivered intravenously at AUC 5 on day 1 every 3 weeks at each dose level of BKM120. Should dose level 3 be completed, carboplatin will be given at AUC 6 and BKM120 at 100 mg.
  In the absence of BKM120 DLT, each level will be administered to 3 patients A minimum of 2 cycles per each dose level will be administered in the absence of disease progression or toxicity
  Other Names: Buparlisib (BKM120); CARBOPLATIN TEVA
  Arms: BKM120-CARBO

SUMMARY:
PI3K signaling is a hallmark of many cancers. Subsets of cancers become dependent on PI3K pathway signaling as a result of mutations of the PIK3CA gene itself or of regulators of PI3K (e.g. PTEN, HER2). As a consequence, pathway mutated tumors are particularly sensitive towards PI3K-pathway inhibition. BKM120 is a potent and highly specific oral pan-class I PI3K-inhibitor.

The study FM-11-F01b is a phase Ib single institution study using the combination of BKM120 and cisplatin or carboplatin in patient with pathologically confirmed recurrent or metastatic advanced solid tumor, for which treatment with a platinum agent is indicated (preferentially head and neck, NSCLC, ovary, endometrial).

The primary objective of the study is to define the phase II recommended dose of daily oral BKM120 and cisplatin (Group 1) or carboplatin (Group 2), given intravenously (IV) on day 1 every 3 weeks.

DETAILED DESCRIPTION:
Despite recent progresses in antineoplastic therapy durable cancer remission is still infrequent in many solid tumors and new treatment options are needed for patients whose cancer has progressed following standard therapies. There is an increasing interest of evaluating new combinations of cytotoxics with new molecule targeted agents which could increase antitumor activity.

PI3K signaling is a hallmark of many cancers. Subsets of cancers become dependent on PI3K pathway signaling as a result of mutations of the PIK3CA gene itself or of regulators of PI3K (e.g. PTEN, HER2). As a consequence, pathway mutated tumors are particularly sensitive towards PI3K-pathway inhibition. BKM120 is a potent and highly specific oral pan-class I PI3K-inhibThe study FM-11-F01b is a phase Ib single institution study using the combination of BKM120 and cisplatin or carboplatin in patient with pathologically confirmed recurrent or metastatic advanced solid tumor, for which treatment with a platinum agent is indicated (preferentially head and neck, NSCLC, ovary, endometrial).

itor. The study treatment foreseen BKM120 administered on a continuous once daily dosing schedule at a dose of 60, 80 or 100 mg (p.o.) plus Carboplatin or Cisplatin. Cisplatin 75 mg/mq will be administered as a 2 hours intravenous infusion every 3 weeks. Carboplatin AUC 5 (or AUC 6 if dose level 3 has been completed) will be administered as a 30 minutes intravenous infusion diluted in 250 mL of normal saline every 3 weeks.

This is a single institution phase I study. Up to 3 dose levels of daily BMK120 will be studied. A standard 3 + 3 phase I dose escalation design will be used for both Group 1 and Group 2. Dose escalation in Group 1 and Group 2 will be mutually independent.

The primary objective of the study is to define the phase II recommended dose of daily oral BKM120 and cisplatin (Group 1) or carboplatin (Group 2), given intravenously (IV) on day 1 every 3 weeks. BKM120 and carboplatin or cisplatin.

ELIGIBILITY:
Inclusion criteria:

* Patient has provided a signed Informed Consent Form (ICF) obtained prior to any screening procedure;
* Patient is ≥ 18 years at the day of consenting to the study
* Patient has an ECOG performance status ≤ 1
* Pathologically confirmed recurrent or metastatic advanced solid tumor, for which treatment with a platinum agent is indicated
* Life expectancy ≥ 6 months
* Patient has adequate bone marrow and organ function
* Patient must be able to swallow and retain oral medication
* Patient may have received more than 1 prior cytotoxic chemotherapy regimens for recurrent or metastatic disease
* Negative serum pregnancy test within 48 hours before starting study treatment in women with childbearing potential
* Patients may receive concurrent radiation therapy to painful bone metastases or areas of impending bone fracture
* Patients must be disease-free of other prior invasive cancers for > 5 year
* Patients must complete all screening assessments as outlined in the protocol

Exclusion Criteria:

* Patient has received previous treatment with PI3K and/or mTOR inhibitors
* Patient has received chemotherapy or targeted anticancer therapy ≤ 4 weeks prior to starting study drug or has not recovered from side effects of such therapy
* Patient has symptomatic CNS metastases (Patients with controlled and asymptomatic CNS metastases may participate in this trial)
* Patient has any of the below mood disorders as judged by the Investigator or a Psychiatrist, or meets the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9)
* Patient is concurrently using other approved or investigational antineoplastic agent
* Patient has received wide field radiotherapy ≤ 4 weeks prior to starting study drug
* Patient has had major surgery within 2 weeks days prior to starting study drug;
* Patients with diabetes mellitus or steroid-induced diabetes mellitus or known intolerance to glucides or fasting glucose > 120 mg/dL or HbA1c > 8 %
* Patient has important cardiac disease

  * LVEF < 50%; NYHA Class III or IV
  * QTc > 480 msec; Congenital long QT syndrome
  * Clinically significant resting bradycardia
  * Complete left bundle branch block; Right bundle branch block + left anterior hemiblock
* Patient has impairment of GI function or GI disease
* Patient receiving chronic treatment with steroids or another immunosuppressive agent.
* Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate his/her participation in the clinical study (e.g.,chronic pancreatitis, active or chronic liver disease, renal disease etc.)
* Patient has diarrhea ≥ 2 CTCAE grade 2
* Preexisting peripheral neuropathy > grade 1
* Patient has been treated with any hematopoietic colony-stimulating growth factors ≤ 2 weeks prior to starting study drug
* Prior hypersensitivity reaction to carboplatin or cisplatin
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or patient has a history of non-compliance to medical regimen
* Patient is currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Patient has a known history of HIV (infection; 21. Patient is a pregnant or nursing (lactating) woman
* Patient is a man or woman of childbearing potential unwilling to use a double barrier method for birth control throughout the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-12; Primary Completion 2017-06-09 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities in each of the study dose levels | 36 months
  Determination of phase II recommended dose of daily oral BKM120 and cisplatin (Group 1) or carboplatin (Group 2), based upon drug related Dose Limiting Toxicities as described in the protocol at the end of Cycle 1 (each cycle is 22 days)

SECONDARY OUTCOMES:
Response rate | 36 months
  Defined as the percentage of complete or partial responders assessed by RECIST criteria (v1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gianni, MD, Study Chair — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No